CLINICAL TRIAL: NCT03366038
Title: Shark Mouth Modified Pancreaticojejunostomy in Pancreaticoduodenectomy Procedure
Brief Title: Shark Mouth Modified Pancreaticojejunostomy
Acronym: SMMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dianrong Xiu, Chief of General Surgery Department, Peking University Third Hospital
Other Study IDs: PekingUTHGS
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer; Periampullary Carcinoma
Keywords: pancreaticoduodenectomy; pancreaticojejunostomy; pancreatic fistula
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Modified Pancreaticojejunostomy: Shark Mouth Modified Pancreaticojejunostomy is performed following pancreaticoduodenectomy.
  Interventions: Procedure: Shark Mouth Modified Pancreaticojejunostomy

INTERVENTIONS:
Procedure: Shark Mouth Modified Pancreaticojejunostomy — The remnant of jejunum is closed by continuous suture. The transverse incision is made on the posterior wall of the jejunum (5 centimeters distal to remnant）, which starts at 0.2 centimeter to the mesenteric border and should never exceed the anti-mesenteric border . In case of large pancreas remnant, a longitudinal jejunum incision will be done at anterior part of anastomosis.
  The posterior part of anastomosis is two layers of intermittent suture, including seromuscular suture layer and full thickness suture layer. The anterior part of anastomosis is a single layer full thickness suture. At last, the seromuscular layer of the proximal jejunum is sutured with the anterior pancreatic capsule to cover the anterior part of anastomosis.

SUMMARY:
Pancreaticoduodenectomy (PD) is one of the most complicated surgical procedure and one of the standard treatments for benign and malignant disease of pancreatic head and periampullary region. Improvements in surgical techniques and the perioperative management of patients undergoing PD have reduced the surgical mortality rates to less than 3% in high-volume medical centers. However, the incidence of postoperative complication remains high, which ranges from 30% to 50% and the pancreatic fistula rate ranges from 5% to 40%. The key point of PD is still the enteric reconstruction of pancreatic stump. There were different techniques of enteric reconstruction, including: invagination pancreaticojejunostomy, binding pancreaticojejunostomy, duct-to-mucosa pancreaticojejunostomy, Roux-en-Y pancreaticojejunostomy, and pancreaticogastrostomy and each technique had its advantages and disadvantages. We established a new digestive reconstruction technique named shark mouth modified pancreaticojejunostomy, which had theoretical advantages including easier performed; lower tension and less complication. The shark mouth modified pancreaticojejunostomy is an end-to-end pancreaticojejunostomy procedure which is between invagination pancreaticojejunostomy and binding pancreaticojejunostomy.The remnant of jejunum is shaped as shark mouth and then sutured with the pancreas remnant. After the surgery, the patients will be well followed up. The pancreaticojejunostomy time, post-operation complication, mortality and hospital stay will be documented to study the safety, efficiency and advantage of this new procedure.

DETAILED DESCRIPTION:
A pancreaticoduodenectomy (PD) still remains the curable treatment choice for most of malignant and benign neoplasms of the head of the pancreas and periampullary region. Though the safety of PD has been significantly improved, the post-operative pancreatic fistula (POPF) always is a formidable complication. More and more attention was focused on the different procedure of enteric reconstruction of pancreatic stump, which might be the key point to reduce the POPF.

This is a prospective clinical trial performed in the general surgery department of Peking University Third Hospital. All pancreatic remnants are reconstructed with the method of Shark Mouth Modified Pancreaticojejunostomy. Shark Mouth Modified Pancreaticojejunostomy is performed as standardized procedure and all the detailed data of this procedure is documented, including gland texture, pancreas duct diameter, size of the stent, width of the pancreatic stump and diameter of the jejunum transverse incision. Silicone tube is inserted as internal stents and fixed on the pancreas remnant with non-absorbable sutures. The distal end of the tube should exceed the anastomosis of the common bile duct and jejunum. The same perioperative management strategies are conducted in all patients. Drainages are placed in all patients during the surgeries. Prophylactic somatostatin analogue are used in all cases for 3 days post operations.

Theoretically, the incision of "Shark Mouth" might facilitate the pancreaticojejunostomy especially for the large pancreatic remnant; the feature of anastomosis might reduce the tension of pancreaticojejunostomy, which is important for the healing of anastomosis and might reduce the risk of POPF in the soft pancreas; the characters of anastomosis permits total drainage of pancreatic remnant, which is crucial in the situation of thinner pancreatic ducts.The purpose of this study is to evaluate the new anastomosis called "Shark Mouth Modified Pancreaticojejunostomy", especially the morbidity of POPF.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer or other diseases which need pancreaticoduodenectomy
* Operation-tolerated
* Informed consent

Exclusion Criteria:

* History of abdominal operation
* Pancreaticoduodenectomy is given up during operation
* Patients require to exit from the study anytime
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients in the Department of General Surgery, Peking University Third Hospital who match to the eligibility criteria will be selected and recruited
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-12-09 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
pancreatic fistula | From 3 days after operation until the date of discharge or date of drains removal, whichever came first, assessed up to 90 days
  The determine of pancreatic fistula follows the International Study Group on Pancreatic Fistulas (ISGPF) criteria.

SECONDARY OUTCOMES:
Mortality | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 90 days
  30-day or in-hospital mortality: death from any cause within 30 days after operation or any in-hospital death are considered concerned with the procedure of pancreaticojejunostomy
Morbidity | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days
  any post-operation complications will be recorded and graded according the Clavien-Dindo Classification of Surgical Complications
pancreaticojejunostomy time | From the start of intraoperative transverse incision on the posterior wall of the jejunum to the finishing of shark mouth modified pancreaticojejunostomy .
  The operation time of pancreaticojejunostomy
Hospital stay | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days
  Post-operation hospital stay will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Dainrong, Doctor, Principal Investigator — Department of General Surgery, Peking University Third Hospital
Locations (1):
- Department of General Surgery, Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Stating 12 months after publication
Access Criteria: All the global researchers may get all the individual participant data by sending emai to xiudianrong7320@163.com

REFERENCES:
- [Background] Chen YJ, Lai EC, Lau WY, Chen XP. Enteric reconstruction of pancreatic stump following pancreaticoduodenectomy: a review of the literature. Int J Surg. 2014;12(7):706-11. doi: 10.1016/j.ijsu.2014.05.060. Epub 2014 May 20. PMID 24851718
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Derived] Wang HY, Li MX, Xiu DR. Shark mouth pancreaticojejunostomy: a new enteric reconstruction procedure of pancreatic stump. Chin Med J (Engl). 2019 Jun 5;132(11):1354-1358. doi: 10.1097/CM9.0000000000000219. PMID 30896569

DOCUMENTS (1):
  • Study Protocol (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03366038/Prot_000.pdf